CLINICAL TRIAL: NCT05012137
Title: The Minimum Effective Volume (MEV) of 0.5% Ropivacaine in Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block (SASIS-FICB)
Brief Title: The MEV of 0.5% Ropivacaine in Ultrasound-guided SASIS-FICB
Acronym: SASIS-FICB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SASIS-FICB
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Nerve Block
Keywords: Minimum Effective volume; Ropivacaine; Fascia Iliaca Compartment Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This is a dosing exploratory study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SASIS-FICB (Experimental): All subjects will be enrolled in the experimental group and receive an Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block (SASIS-FICB)
  Interventions: Procedure: Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block (SASIS-FICB) with 0.5% ropivacaine; Drug: different volume of 0.5% ropivacaine

INTERVENTIONS:
Procedure: Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block (SASIS-FICB) with 0.5% ropivacaine — all the patients received Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block (SASIS-FICB)
Drug: different volume of 0.5% ropivacaine — According to the subject's response to the injection dose, the next subject will be injected with a different volume of the drug according to the preset rules

SUMMARY:
The Aim of This Study is to Determine the Minimum Effective Volume of Local Anesthetic (Ropivacaine 0.5%) Required to Produce an Effective Ultrasound-guided Supra-anterior Superior Iliac Spine Fascia Iliaca Compartment Block（SASIS-FICB） for Surgical Anesthesia in 90% of Patients Scheduled for Elective Surgery of One Lower Limbs.

DETAILED DESCRIPTION:
The study is based on biased coin design, and the volume of Local Anesthetic (Ropivacaine 0.5%) for the next patient is determined by the result of the last one. In the case of block failure, the volume will be increased by 2.5ml. Conversely, block success will result in either a reduction in volume by 2.5ml (probability 11%) or no change in volume (probability 89%). A blinded assistant will assess sensory and motor blockade in each nerve territory ( the femoral, obturator and lateral femoral cutaneous nerves) at 5-min intervals up to 30 min after completion of the block. Finally, MEV90 is calculated by isotonic regression.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hip/knee surgery

Exclusion Criteria:

* age <18 years
* body mass index >35
* inability to consent to the study
* allergy to local anesthetics
* a history of liver or renal insufficiency, coagulopathy
* clinical evidence of peripheral neuropathies, abnormalities of sensory or motor function of the FN, ON or LFCN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-08-25 (Estimated); Primary Completion 2021-10-25 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
The MEV90 of 0.5%Ropivacaine in Ultrasound-guided SASIS-FICBS | up to 6 months
  We prospectively recruited patients to receive different volumes of SASIS-FICB in accordance with the sequential trial rules of biased coins until 45 successful SASIS-FICB attempts were completed. MEV90 was calculated by isometric regression.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Study Chair — Director of Anesthesiology Department,Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No